CLINICAL TRIAL: NCT04243278
Title: Postpartum Low-Dose Aspirin After Preeclampsia for Optimization of Cardiovascular Risk (PAPVASC)
Acronym: PAPVASC
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Poor Recruitment Rates
Sponsor: Dr. Graeme Smith (Other)
Responsible Party: Sponsor-Investigator, Dr. Graeme Smith, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: OBGY-43312-20
Record Dates: First submitted 2020-01-09; First posted 2020-01-28 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Preeclampsia Severe; Cardiovascular Diseases; Primary Prevention
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PO LD-ASA (Experimental): Study participants who are assigned to the oral aspirin arm of the study will receive 81mg oral aspirin. Over-encapsulated 81mg aspirin tablets will be used. Study participants in this arm will take 81mg aspirin daily for 6 months.
  Interventions: Drug: Low-dose aspirin
- PO Placebo (Placebo Comparator): A standard placebo pill, the same size, shape and color of the oral aspirin will be used. The placebo pills will be over-encapsulated in the same manner as the aspirin tablets. The placebo will be administered to the participants randomized to placebo group in the same manner the oral aspirin would be administered - they will take the pill daily for 6 months.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Low-dose aspirin — 81 mg of low dose aspirin PO for 6 months
  Arms: PO LD-ASA
Drug: Placebo oral tablet — placebo PO for 6 months
  Arms: PO Placebo

SUMMARY:
Women who develop preeclampsia (PE) in pregnancy are at a greater risk for adverse cardiovascular health outcomes. PE is associated with vascular remodeling and functional changes in the postpartum, reflective of its systemic effects during gestation. Aberrant microvascular endothelial function has been demonstrated in pharmacological studies of formerly preeclamptic women. However, clinicians do not have any recourse for modulating vascular functional adaptations nor mitigating the future risk for maternal disease in the early postpartum. Low-dose aspirin (LD-ASA) is commonly prescribed to prevent PE and confers a consistently positive effect on mitigating PE risk when given in early gestation to women at risk. While the precise effect of LD-ASA on PE development is not fully understood, existing evidence suggests it may confer an array of anti-thrombotic, vasodilatory, pro-endothelial effects that mitigate the risk of disease.

This study will be a randomized, placebo-controlled trial of LD-ASA administration over 6 months in the early postpartum in women with prior severe PE. Women will be identified, enrolled, and randomized to either treatment or placebo groups. Treatment groups will receive 81 mg daily oral aspirin, while control groups will receive an equivalent placebo pill. Vascular functional assessment at study outset will take place, combining laser speckle contrast imaging and iontophoresis of dilute vasoactive drug solutions. Blood and urine will be obtained for analysis of cardiometabolic and endothelial factors. Participants will take their assigned study drug for 6 months, after which a retest appointment will take place to assess vascular functional changes.

DETAILED DESCRIPTION:
This study will be a prospective, randomized, controlled, double-blinded, single-centre trial with two parallel groups. The primary outcome will be endothelium-dependent vasodilation as measured by iontophoresis and laser speckle contrast imaging (LSCI).

Participants will be recruited following a preeclamptic delivery at Kingston Health Sciences Center. Following confirmation of eligibility, they will be randomized to treatment or control groups. Randomization will be performed as block randomization with a 1:1 allocation ratio. In total, 44 participants will be recruited and randomized, with 22 being assigned to each treatment arm.

Prior to discharge from the hospital, investigators will assess both vascular functional and biochemical variables in each participant. Using LSCI, a non-invasive imaging modality, investigators will continuously measure microvascular blood flow in the volar forearm in response to dilute drug solutions administered using iontophoresis. Iontophoresis refers to the non-invasive administration of drugs under the influence of an applied current. Iontophoresis of acetylcholine, an endothelium-dependent vasodilator, and sodium nitroprusside, an endothelium-independent vasodilator, will occur, the response to which will be recorded using LSCI.

At the study outset, investigators will record additional biophysical parameters such as blood pressure, weight, and BMI. Blood will be drawn and serum analysis of lipid profile, fasting glucose, high sensitivity C-reactive protein, s-Flt-1, platelet-derived growth factor, and uric acid will occur. Urine will be collected for analysis of albumin: creatinine ratio. Findings will then be integrated to calculate a lifetime cardiovascular risk score, which is used to categorize individuals as low risk or high risk.

Study participants who are assigned to the oral aspirin arm of the study will receive 81 mg oral aspirin. Over-encapsulated 81mg aspirin tablets will be used. Study participants in this arm will take 81mg aspirin daily for 6 months. A standard placebo pill, the same size, shape, and color of the oral aspirin will also be used. The placebo will be administered to the participants randomized to the placebo group in the same manner the oral aspirin would be administered - they will take the pill daily for 6 months.

On a monthly basis, all participants will be contacted by study personnel to confirm that they have been taking their medication, and that there are no adverse effects to report.

In addition to either LD-ASA or placebo, both groups will receive our center's current standard of care of cardiovascular assessment and lifestyle counseling at the Maternal Health Clinic (MHC) at Kingston Health Sciences Center. MHC appointments take place at 6 months postpartum. At the MHC appointment, vascular reactivity testing will occur again, followed by biochemical analyses, to assess vascular functional recovery due to the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed severe preeclampsia diagnosed prior to delivery

   Preeclampsia defined as: Blood pressure > 140/90 AND proteinuria > 300mg/24 hours OR 2+ on repeat dip stick

   Severe Preeclampsia defined as the presence of one or more of the following:

   i. systolic blood pressure ≥ 160mmHg or diastolic blood pressure ≥ 110 mmHg on 2 occasions at least 4 hours apart

   ii. new-onset cerebral or visual disturbance

   iii. severe persistent right upper quadrant pain or serum transaminase concentrations ≥ 2 times the upper limit of normal

   iv. thrombocytopenia (platelets < 100 x 109/L)

   v. renal insufficiency (serum creatinine > 97.2 umol/L)

   vi. pulmonary edema
2. A singleton gestation
3. Gestation between 24+0/7 to 40+6/7 weeks.Exclusion Criteria:

Exclusion Criteria:

1. Multiple pregnancy
2. Chronic hypertension or other condition requiring the use of BP-lowering medication
3. Cardiovascular disorders: Unstable angina pectoris, heart failure, life-threatening arrhythmia, atrial fibrillation, kidney failure
4. Known allergy or sensitivity to aspirin used in the study
5. Any medical comorbidity that is a contraindication to LD-ASA: Hemophilia or other bleeding disorder, history of GI bleeding, renal failure, severe liver disease, thrombocytopenia, gout, G6PD deficiency
6. Recent history of drug/alcohol abuse (< 1 year prior to delivery), or receiving treatment for such
7. Nasal polyps
8. Hypercholesterolemia requiring pharmaceutical treatment
9. Raynaud's phenomenon
10. Collagen-vascular disease: lupus, scleroderma, rheumatoid arthritis
11. History of pre-existing diabetes
12. Ongoing use of any of the following medications: methotrexate, anti-coagulants, thrombolytics, oral hypoglycemics, uricsuric agents, valproic acid, glucocorticosteroids, digoxin

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Endothelium-Dependent Dilation | Immediate Postpartum to 6 Months Postpartum
  Changes in endothelium-dependent dilation from the immediate postpartum period to 6 months postpartum. Measured by laser speckle contrast imaging in conjunction with iontophoresis.

SECONDARY OUTCOMES:
Endothelium-Independent dilation | Immediate Postpartum to 6 Months Postpartum
  Changes in endothelium-independent dilation from the immediate postpartum period to 6 months postpartum. Measured by laser speckle contrast imaging in conjunction with iontophoresis.
Blood Pressure | 6 months postpartum
  Blood pressure will be taken as the average of five consecutive measurements using an automated controller (BPTru).
Body Mass Index | 6 months postpartum
  Height and weight will be measured at 6 months postpartum and body mass index will be calculated.
Concentration of Serum sFlt-1 | 6 months postpartum
  A serum blood sample will be taken and sFlt-1 levels will be analysed in our basic science lab.
Concentration of Placental Growth Factor | 6 months postpartum
  A serum blood sample will be taken and placental growth factor levels will be analysed in our basic science lab.
High Sensitivity C-Reactive Protein | 6 months postpartum
  A serum blood sample will be sent to our hospital lab. A clinical level of high sensitivity c-reactive protein will be measured.
Uric Acid Levels | 6 months postpartum
  A serum blood sample will be sent to our hospital lab. A clinical level of uric acid will be measured.
Total Cholesterol | 6 months postpartum
  A serum blood sample will be sent to our hospital lab. A clinical lipid profile will be measured, including total cholesterol.
High Density Lipoprotein | 6 months postpartum
  A serum blood sample will be sent to our hospital lab. A clinical lipid profile will be measured, including high density lipoprotein.
Low Density Lipoprotein | 6 months postpartum
  A serum blood sample will be sent to our hospital lab. A clinical lipid profile will be measured, including low density lipoprotein.
Triglycerides | 6 months postpartum
  A serum blood sample will be sent to our hospital lab. A clinical lipid profile will be measured, including triglycerides.
Urine Albumin Creatinine Ratio | 6 months postpartum
  A urine sample will be collected and sent to our hospital lab. A clinical urine albumin creatinine ratio will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Graeme N Smith, MD, PhD, Principal Investigator — Queen's Department of Obstetrics and Gynaecology
Locations (1):
- Queen's University Department of Obstetrics and Gynecology, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No